CLINICAL TRIAL: NCT00694356
Title: A Phase I Study of MK-0646 in Patients With Relapsed or Refractory Locally Advanced or Metastatic Solid Tumors
Brief Title: Study of Dalotuzumab (MK-0646) in Adults With Solid Tumors (MK-0646-009)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0646-009; 2008_012 (Other: Telerex Study Number)
Record Dates: First submitted 2008-05-29; First posted 2008-06-10 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-07

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — dalotuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dalotuzumab 5 mg/kg (Experimental): Participants receive dalotuzumab 5 mg/kg by intravenous (IV) infusion once each week for up to 1 year or until participant withdraws consent, experiences an adverse event (AE), progressive disease or major protocol violation, has moved or is lost to follow up.
  Interventions: Biological: Dalotuzumab
- Dalotuzumab 10 mg/kg (Experimental): Participants receive dalotuzumab 10 mg/kg by IV infusion once each week for up to 1 year or until participant withdraws consent, experiences an AE, progressive disease or major protocol violation, has moved or is lost to follow up.
  Interventions: Biological: Dalotuzumab
- Dalotuzumab 15 mg/kg/7.5 mg/kg (Experimental): Participants receive an initial dose of dalotuzumab 15 mg/kg by IV infusion followed by a maintenance dose of dalotuzumab 7.5 mg/kg by IV infusion once every 2 weeks for up to 1 year or until participant withdraws consent, experiences an AE, progressive disease or major protocol violation, has moved or is lost to follow up.
  Interventions: Biological: Dalotuzumab

INTERVENTIONS:
Biological: Dalotuzumab — IV infusion
  Other Names: MK-0646

SUMMARY:
This clinical study evaluates the safety, tolerability, pharmacokinetics, and immunogenicity of dalotuzumab (MK-0646) in participants with relapsed or refractory locally advanced or metastatic solid tumors using once weekly and once every other week dose infusion regimens.

The primary study hypothesis is that administration of dalotuzumab as a once weekly and an every other week infusion will be generally safe and well tolerated

ELIGIBILITY:
Inclusion Criteria:

* Has histologically- or cytologically-confirmed metastatic or locally advanced solid tumor(s) that has (have) failed to respond to standard therapy, or for which adequate standard therapy does not exist
* Has tumor(s) associated with insulin-like growth factor 1 receptor (IGF-1R) expression in the literature (e.g. prostate, pancreatic, colon, lung and breast)
* Has Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Demonstrates adequate organ function

Exclusion Criteria:

* Has had chemotherapy, radiotherapy, or biological therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to registration
* Is concurrently using growth hormone (GH), or growth hormone inhibitor
* Has any active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has any primary CNS tumor - any symptomatic ascites or plural effusion
* Has a history or current evidence of any clinically significant disease that might confound the results of the study, complicate the interpretation of the study results, interfere with the participant's participation, or pose an additional risk to the participant
* Is pregnant or breast-feeding

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-08-04 (Actual); Primary Completion 2009-03-18 (Actual); Study Completion 2009-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dalotuzumab 5 mg/kg | Dalotuzumab 10 mg/kg | Dalotuzumab 15 mg/kg/7.5 mg/kg
Started | 3 | 6 | 6
Completed | 0 | 0 | 0
Not Completed | 3 | 6 | 6
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Progressive Disease | 2 | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Dalotuzumab 5 mg/kg: Participants receive dalotuzumab 5 mg/kg by IV infusion once each week for up to 1 year or until participant withdraws consent, experiences an AE, progressive disease or major protocol violation, has moved or is lost to follow up.
- Total: Total of all reporting groups
Arm/Group | Dalotuzumab 5 mg/kg | Dalotuzumab 10 mg/kg | Dalotuzumab 15 mg/kg/7.5 mg/kg | Total
Number analyzed (Participants) | 3 | 6 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.3 (1.5) | 63.5 (3.9) | 59.2 (14.2) | 62.3 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 4
  Male | 3 | 4 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced a Dose-limiting Toxicity (DLT)
Description: Toxicity was graded and recorded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. DLTs were defined as the occurrence of any of the following events when judged to be related to the study medication: Grade 4 neutropenia; Grade 3 neutropenia with fever >38.5°C; Grade 4 thrombocytopenia; Grade 3 or Grade 4 non-hematologic toxicity, except alopecia and inadequately treated diarrhea, nausea and vomiting. The number of participants who experienced a DLT is presented.
Time Frame: Cycle 1 (Up to 4 weeks)
Population: The population consisted of all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Dalotuzumab 5 mg/kg | Dalotuzumab 10 mg/kg | Dalotuzumab 15 mg/kg/7.5 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study treatment, whether or not considered related to the use of study treatment. Any worsening (i.e. any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which was temporally associated with the use of study treatment, was also an AE. The number of participants who experienced at least one AE is presented.
Time Frame: Up to 30 days after last dose of study treatment (Up to 101 days)
Population: The population consisted of all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Dalotuzumab 5 mg/kg | Dalotuzumab 10 mg/kg | Dalotuzumab 15 mg/kg/7.5 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
Participants | 3 | 6 | 6

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an AE
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the study treatment, whether or not considered related to the use of study treatment. Any worsening (i.e. any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition which was temporally associated with the use of study treatment, was also an AE. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to 71 days
Population: The population consisted of all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Dalotuzumab 5 mg/kg | Dalotuzumab 10 mg/kg | Dalotuzumab 15 mg/kg/7.5 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
Participants | 1 | 0 | 0

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Dalotuzumab
Description: Cmax was assessed on Week 2 (Day 8) for the Dalotuzumab 5 mg/kg and Dalotuzumab 10 mg/kg treatment groups and on Week 3 (Day 15) for the Dalotuzumab 15 mg/kg/7.5 mg/kg treatment group.
Time Frame: Pre-dose, 0.5 h after start of infusion, end of infusion, 5, 10, 24, 30, 48 and 96 and 168 h post-dose
Population: The population consisted of all participants who had pharmacokinetic (PK) measurements at Baseline and at least once during treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Dalotuzumab 5 mg/kg | Dalotuzumab 10 mg/kg | Dalotuzumab 15 mg/kg/7.5 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
µg/mL | 85.60 (6.94) | 161.78 (23.02) | 244.05 (11.57)

5. Secondary Outcome: Area Under the Concentration-Time Curve From Zero to Infinity (AUC0-∞) of Dalotuzumab
Description: AUC0-∞ was assessed on Week 2 (Day 8) for the Dalotuzumab 5 mg/kg and Dalotuzumab 10 mg/kg treatment groups and on Week 3 (Day 15) for the Dalotuzumab 15 mg/kg/7.5 mg/kg treatment group.
Time Frame: Pre-dose, 0.5 h after start of infusion, end of infusion, 5, 10, 24, 30, 48 and 96 and 168 h post-dose
Population: The population consisted of all participants who had PK measurements at Baseline and at least once during treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/mL
Arm/Group | Dalotuzumab 5 mg/kg | Dalotuzumab 10 mg/kg | Dalotuzumab 15 mg/kg/7.5 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
mg*h/mL | 11.72 (10.06) [1.0 to 1.0] | 21.71 (37.64) [1.0 to 5.0] | 38.99 (21.27) [1.0 to 1.0]

6. Secondary Outcome: Time to Cmax (Tmax) of Dalotuzumab
Description: Tmax was assessed on Week 2 (Day 8) for the Dalotuzumab 5 mg/kg and Dalotuzumab 10 mg/kg treatment groups and on Week 3 (Day 15) for the Dalotuzumab 15 mg/kg/7.5 mg/kg treatment group.
Time Frame: Pre-dose, 0.5 h after start of infusion, end of infusion, 5, 10, 24, 30, 48 and 96 and 168 h post-dose
Population: The population consisted of all participants who had PK measurements at Baseline and at least once during treatment.
Measure: Median (Full Range); unit: h
Arm/Group | Dalotuzumab 5 mg/kg | Dalotuzumab 10 mg/kg | Dalotuzumab 15 mg/kg/7.5 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
h | 1.0 (1.0) [1.0 to 1.0] | 3.0 (23.02) [1.0 to 5.0] | 1.0 (11.57) [1.0 to 1.0]

7. Secondary Outcome: Apparent Terminal Half-life (t1/2) of Dalotuzumab
Description: t1/2 was assessed on Week 2 (Day 8) for the Dalotuzumab 5 mg/kg and Dalotuzumab 10 mg/kg treatment groups and on Week 3 (Day 15) for the Dalotuzumab 15 mg/kg/7.5 mg/kg treatment group.
Time Frame: Pre-dose, 0.5 h after start of infusion, end of infusion, 5, 10, 24, 30, 48 and 96 and 168 h post-dose
Population: The population consisted of all participants who had PK measurements at Baseline and at least once during treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Dalotuzumab 5 mg/kg | Dalotuzumab 10 mg/kg | Dalotuzumab 15 mg/kg/7.5 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
h | 129.85 (12.44) [1.0 to 1.0] | 110.36 (20.18) [1.0 to 5.0] | 167.09 (20.94) [1.0 to 1.0]

8. Secondary Outcome: Clearance (CL) of Dalotuzumab
Description: CL of dalotuzumab was assessed on Week 2 (Day 8) for the Dalotuzumab 5 mg/kg and Dalotuzumab 10 mg/kg treatment groups and on Week 3 (Day 15) for the Dalotuzumab 15 mg/kg/7.5 mg/kg treatment group.
Time Frame: Pre-dose, 0.5 h after start of infusion, end of infusion, 5, 10, 24, 30, 48 and 96 and 168 h post-dose
Population: The population consisted of all participants who had PK measurements at Baseline and at least once during treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min/kg
Arm/Group | Dalotuzumab 5 mg/kg | Dalotuzumab 10 mg/kg | Dalotuzumab 15 mg/kg/7.5 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
mL/min/kg | 0.0071 (10.06) | 0.0077 (37.64) | 0.0064 (21.27)

9. Secondary Outcome: Steady State Volume of Distribution (Vss) of Dalotuzumab
Description: Vss was assessed on Week 2 (Day 8) for the Dalotuzumab 5 mg/kg and Dalotuzumab 10 mg/kg treatment groups and on Week 3 (Day 15) for the Dalotuzumab 15 mg/kg/7.5 mg/kg treatment group.
Time Frame: Pre-dose, 0.5 h after start of infusion, end of infusion, 5, 10, 24, 30, 48 and 96 and 168 h post-dose
Population: The population consisted of all participants who had PK measurements at Baseline and at least once during treatment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/kg
Arm/Group | Dalotuzumab 5 mg/kg | Dalotuzumab 10 mg/kg | Dalotuzumab 15 mg/kg/7.5 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
L/kg | 0.0776 (17.46) | 0.0740 (24.10) | 0.0924 (16.74)

10. Secondary Outcome: Number of Participants Who Developed a Human Anti-Humanized Antibody (HAHA) Response to Dalotuzumab
Description: Formation of HAHAs may block efficacy by substantially increasing the clearance of dalotuzumab and limit the possibility of future dalotuzumab therapy. The occurrence of HAHAs in the sera of dalotuzumab treated participants at any of the serum collection times was assessed.
Time Frame: Cycle 1: predose on Days 1, 8, 15, and 22; Cycles 2 and 3: predose on Day 1; 4 weeks after last dose of study drug
Population: The population consisted of all participants who received at least one dose of study treatment.
Measure: Number; unit: Participants
Arm/Group | Dalotuzumab 5 mg/kg | Dalotuzumab 10 mg/kg | Dalotuzumab 15 mg/kg/7.5 mg/kg
Number analyzed (Participants) | 3 | 6 | 6
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of study treatment (Up to 101 days)
Description: The population consisted of all participants who received at least one dose of study treatment.
Arm/Group | Dalotuzumab 5 mg/kg | Dalotuzumab 10 mg/kg | Dalotuzumab 15 mg/kg/7.5 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalotuzumab 5 mg/kg (N=3) | Dalotuzumab 10 mg/kg (N=6) | Dalotuzumab 15 mg/kg/7.5 mg/kg (N=6)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dalotuzumab 5 mg/kg (N=3) | Dalotuzumab 10 mg/kg (N=6) | Dalotuzumab 15 mg/kg/7.5 mg/kg (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Fatigue (General disorders) | 1 (1) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time shortened (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 4 (4) | 1 (1)
Blood urea increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
International normalised ratio decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Prothrombin time shortened (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 2 (2) | 3 (3)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (6) | 4 (5)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Ketonuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 1 (3) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.